CLINICAL TRIAL: NCT00510640
Title: Phase 2 of Sunitinib (Sutent) in Patients With Locally Advanced or Metastatic Anaplastic, Differentiated or Medullar Thyroid Cancer
Brief Title: Thyroid Cancer and Sunitinib
Acronym: THYSU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9277-06; 2006-23
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Cancer; Thyroid Carcinoma
Keywords: thyroid carcinoma; Sunitinib; RECIST guidelines
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Sunitinib will be administered orally daily for 4 weeks followed by a 2-week rest; the daily starting dose will be 50 mg with a provision for dose reduction based on tolerability. All patients will receive repeated cycles until disease progression or occurrence of severe toxicity.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Capsule, 12.5 or 50 mg, starting dose level 50 mg daily

SUMMARY:
Due to arguments showing that angiogenesis could be involved in progression of metastatic thyroid carcinoma and to objective response during previous studies with sunitinib (an angiogenic oncology drug also known as Sutent), this study, THYSU, is justified to evaluate the efficacy of sunitinib in metastatic thyroid carcinoma. Furthermore, the standard treatment of metastatic thyroid carcinoma when a general treatment is to be prescribed is limited to radioiodine. When radioiodine becomes ineffective, there is no standard treatment despite some use of chemotherapy.

The objective of the trial is to determine the objective tumor response rate (efficacy) in patients with locally advanced or metastatic anaplastic, differentiated or medullary thyroid carcinoma treated with sunitinib; a secondary objective is to evaluate the safety of sunitinib in these patients.

The THYSU trial is a phase II, French multi-center study. This trial's plan is to enroll 75 patients with locally advanced or metastatic anaplastic, differentiated or medullar thyroid carcinoma.

DETAILED DESCRIPTION:
The THYSU trial is a phase II trial of sunitinib (Sutent) in patients with locally advanced or metastatic anaplastic, differentiated or medullary thyroid carcinoma.

Due to arguments showing that angiogenesis could be involved in progression of metastatic thyroid carcinoma and to objective response during a phase I trial with sunitinib, it was justified to evaluate in a prospective trial the efficacy of sunitinib in metastatic thyroid carcinoma. Furthermore, the standard treatment of metastatic thyroid carcinoma when a general treatment is to be prescribed is limited to radioiodine. When radioiodine becomes ineffective, there is no standard treatment despite some usage of chemotherapy.

The objective of the trial is to determine the objective tumor response rate in patients with locally advanced or metastatic anaplastic, differentiated or medullary thyroid carcinoma treated with sunitinib, a secondary objective is to evaluate the safety of sunitinib in these patients with thyroid carcinoma.

The treatment of sunitinib is the standard dosage and schedule. Sunitinib is given orally at the dose of 50 mg daily for 28 days followed by 2 weeks of rest. Forthcoming cycles remain identical. Modification of the dose may use a lower dose at 37.5 mg or 25 mg given daily on the same schedule. All patients will receive repeated cycles of treatment until disease progression, occurrence of unacceptable toxicity, withdrawal of patient consent, or other withdrawal criteria are met. After discontinuation of treatment and the mandated 28-day follow up, patients will be followed only in order to collect information on further antineoplastic therapy and survival. In patients discontinuing treatment for reasons other than disease progression, tumor assessment will continue until disease progression, or initiation of other antineoplastic therapies.

The more frequent side effects are asthenia, mucositis, arterial hypertension, hand foot syndrome and diarrhea. Other side effects have been reported including nausea, vomiting, cutaneous events, decrease in left ventricular ejection fraction, neutropenia, and thrombopenia.

The patients must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

* Patients must sign and date IRB/EC-approved informed consent.
* Age ≥ 18.
* Patients must have a life expectancy of at least 3 months and Karnofsky performance status ≥ 70%
* Patients must have histologically confirmed TC
* Tumor disease must be progressive (evidence of disease progression within 6 months)
* Patients should not be candidates for surgical resection, external beam radiotherapy or radioiodine, and patients must not have more than one previous systemic treatment for cancer
* Patients must have measurable disease defined by RECIST criteria as at least one lesion at least 2 cm in length by conventional CT techniques or at least 1 cm by spiral CT scan.
* Resolution of all acute toxic effects of any prior treatment to NCI - CTCAE (version 3.0) grade < 1.
* Patients must have discontinued from radiation therapy at least 4 weeks before first dose of study treatment and must have recovered from any toxic effects of treatment.
* Blood pressure < 140 / 90 mmHg
* Patients must have adequate organ function.
* Patients with reproductive potential must use medically acceptable contraceptive method.
* Willingness and ability to comply with the study procedures.
* Patient affiliated with or profiting from a social security system

The presence of any non-inclusion criteria will exclude a patient from study enrollment.

Prior to undergoing any specific study procedures, patient and investigator sign informed consent. During the initial visit including verification of eligibility criteria, an interview with the patient is conducted regarding his/her recent and past clinical and treatment history (including oncology history). Physical examination including examination of major body systems, Karnofsky performance status, body weight, height, and vital signs is performed. Laboratory data are collected (hematology and chemistry, coagulation, thyroid tests, tumor markers and pregnancy test if applicable). Para clinic evaluations (12-lead ECGs and tumor imaging) are carried out. LVEF assessed by Echocardiogram or by MUGA scan (if necessary) and Brain Naturatic Peptide (Or NT pro-BNP) test are done.

During the follow-up, the patients are followed between the end of week 4 and week 6 by clinical and biological evaluation. Evaluation of tumor sites under sunitinib is planned every 2 cycles with CT scans. For patients with anaplastic or differentiated thyroid carcinoma, the first stage will include 21 efficacy-evaluable patients. An additional 29 efficacy-evaluable patients will be included at the second stage.

For patients with medullary thyroid carcinoma, the first stage will include 11 efficacy-evaluable patients. An additional 7 to 14 efficacy-evaluable patients will be included at the second stage.

10 French Oncology Departments are involved in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥ 18.
* Patients must have a life expectancy of at least 3 months
* Patients must have a Karnofsky performance status ≥ 70%
* Patients must have histologically confirmed thyroid cancer (TC)
* Tumor disease must be progressive (evidence of disease progression within 6 months before starting the study for follicular and medullary thyroid cancer or symptomatic disease)
* Patients should not be candidates for surgical resection, external beam radiotherapy or radioiodine
* Patients must have measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST), such as at least one lesion at least 2 cm in length by conventional computed tomography (CT) techniques or at least 1 cm by spiral CT scan
* Patients must not have more than one previous systemic treatment for cancer
* Resolution of all acute toxic effects of any prior local treatment to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 3.0) grade < 1
* Patients must have discontinued from radiation therapy at least 4 weeks before start of study treatment and must have recovered from any toxic effects of treatment
* Blood pressure < 140 / 90 mmHg
* Patients must have adequate organ function defined as: Platelets > 100 x 10*9/L, Hemoglobin > 8 g/dl, ANC > 1.5 x 10*9/L, Bilirubin < 3 mg/dL, AST and ALT < 2.5 x the upper limit of normal (ULN) or < 5 x the ULN for liver metastases, INR < 1.7 or prothrombin time < 6 sec over ULN, Serum creatinine < 1.5 x ULN
* Patients with reproductive potential must use medically acceptable contraceptive methods (oral contraception or an intrauterine device [IUD])
* Willingness and ability to comply with all study procedures
* Affiliated or profit patient of a social security system

Exclusion Criteria:

* Prior treatment on sunitinib or other anti-angiogenic therapy
* NCI CTCAE grade 3 hemorrhage < 4 weeks of starting study treatment
* Diagnosis of any second malignancy < 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix uteri that has been adequately treated with no evidence of recurrent disease for 12 months
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
* Any of the following within the 12 months prior to study drug administration: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, including transient ischemic attack, or pulmonary embolism
* Ongoing cardiac dysrhythmias of NCI CTCAE grade > 2, atrial fibrillation of any grade, or prolongation of the QTc interval to > 450 msec for males or > 470 msec for females
* Left ventricular ejection fraction ( LVEF) < 50%
* Hypertension that cannot be controlled by medications
* Treatment with anticoagulant agents and treatment with therapeutic doses of warfarin currently or within 2 weeks prior to first day of sunitinib administration
* Inability to swallow oral medications, or presence of active inflammatory bowel disease, partial or complete bowel obstruction or chronic diarrhea
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
* Pregnancy or breastfeeding
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Receipt of any investigational agent prior to study entry
* Current treatment on another therapeutic clinical trial
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) : defined as the proportion of patients with confirmed complete (CR) or partial response (PR) according to the RECIST, relative to the total patients enrolled who received at least 1 dose of trial medication | Every two cycles

SECONDARY OUTCOMES:
Evaluate the safety of sunitinib in patients with thyroid carcinoma | After each cycle of treatment
Determine time-to-event variables of overall survival, time to: disease progression, response, and duration of response | variable

CONTACTS AND LOCATIONS:
Overall Officials: Alain Ravaud, Pr., Principal Investigator — University Hospital, Bordeaux, France; Geneviève Chene, Pr., Study Chair — University Hospital, Bordeaux, France
Locations (15):
- France (15):
  - Centre Paul Papin - 2 rue Moll, Angers
  - Département Endocrinolo-Diabéto-Nutrition - CHU d'Angers - 4 rue de Larray, Angers
  - Service d'Oncologie Médicale et de Radiothérapie - Hôpital Saint André - 1 rue Jean Burguet, Bordeaux
  - Fédération Endocrinologie - Groupe Hospitalier Est - Hôpital neurologique - CHU Lyon - 59 Boulevard Pinel, Bron
  - Service d'Endocrinologie et maladies métaboliques, Clinique Marc Linquette - rue du Pr Laguesse, Lille
  - Centre Léon Bérard - Département de Médecine - 28 rue Laennec, Lyon
  - Service d'Endocrinologie, CHU Timone, AP-HM - 254 rue St Pierre, Marseille
  - Service des Maladies Endocriniennes - Hôpital Lapeyronie - 191 avenue du Doyen Gaston Giraud, Montpellier
  - Centre Paul Lamarque - Va d'Aurelle - CRLC Val d'Aurelle - 208 rue des Apothicaires, Montpellier
  - Centre Antoine Lacassagne - 33 avenue de Valombrose, Nice
  - Service d'Endocrinologie - Hôpital de l'Archet I - Route Saint Antoine de Jinestière, Nice
  - Service de Cancérologie Médicale - HEGP - 20 rue Leblanc, Paris
  - Service d'Oncologie Médicale, Institut Claudius Regaud - 20-24 rue du Pont Saint Pierre, Toulouse
  - Service d'endocrinologie et Maladies Métaboliques, Groupe Hospitalier Rangueil-Larrey CHU Toulouse - avenue Prof Jean Poulhes, Toulouse
  - Service d'Endocrinologie - CHU de Nancy, Hôpital de Brabois - rue du Morvan, Vandœuvre-lès-Nancy